CLINICAL TRIAL: NCT05774275
Title: A Prospective Phase Ib/II Trial of Preoperative Radiotherapy Combined With Chemotherapy and Immunotherapy in High-Risk Localized Soft Tissue Sarcoma
Brief Title: The Combination of Radiotherapy, Chemotherapy and Immunotherapy in High-Risk Localized Soft Tissue Sarcoma
Acronym: RAPID
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2021-373-2676
Record Dates: First submitted 2023-02-02; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: High-Risk Localized Soft Tissue Sarcoma
MeSH Terms: interventions — liposomal doxorubicin; Doxorubicin; spartalizumab; sintilimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): There will be 52 patients with high-risk localized extremity and trunk soft tissue sarcoma recruited.
  In safety lead-in phase (phase Ib): using 3+3 design, patients will receive 4 cycles of Doxil or doxorubicin hydrochloride, sintilimab and radiotherapy.
  In phase II: Doxil in RP2D, sintilimab and radiotherapy will be applied as before.
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Doxorubicin; Drug: Anti-PD-1 monoclonal antibody; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — In phase Ib: 37.5 mg/m2, 30 mg/m2, d1, q3w; In phase II: recommended phase 2 dose (RP2D), d1, q3w.
  Other Names: Doxil
Drug: Doxorubicin — 75mg/m2, d1, q3w Doxorubicin hydrochloride will be administered if subject is allergic to Doxil.
  Other Names: Doxorubicin Hydrochloride
Drug: Anti-PD-1 monoclonal antibody — 200 mg, d1, q3w
  Other Names: Sintilimab
Radiation: Radiotherapy — BED=50-60Gy(α/β=10); Radiation dose depends on tumor characteristics and organs at risk.

SUMMARY:
This is a prospective, single-center, single-arm, phase Ib/II clinical trial. The study aims to evaluate the safety and efficacy of the treatment which combines radiotherapy, chemotherapy and immunotherapy in patients with high-risk localized soft tissue sarcoma.

There will be 52 patients with high-risk localized extremity and trunk soft tissue sarcoma recruited. The trail is designed as a two-stage study. In safety lead-in phase (phase Ib), using 3+3 design, 4 cycles of Doxil (37.5 mg/m2, 30 mg/m2, q3w) or doxorubicin hydrochloride (75mg/m2, q3w), Sintilimab (200mg, q3w) and radiotherapy (BED=50-60Gy (α/β=10)) will be applied. In phase II, Doxil will be applied in the recommended phase 2 dose (RP2D) according to phase Ib. And 200mg sintilimab and radiotherapy will be applied as before. The dose-limiting toxicity (DLT) in phase Ib and objective response rate (ORR) in phase Ib+Phase II will be mainly analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed STS, G2 or G3. The histological types include: pleomorphic undifferentiated sarcoma, liposarcoma, leiomyosarcoma, synovial sarcoma, myxofibrosarcoma, fibrosarcoma, angiosarcoma but not radiotherapy-induced angiosarcoma, etc.
2. Has>5 cm lesions, or the lesions are determined to be borderline resectable or unresectable by a multidisciplinary consultation.
3. Has imaging-confirmed localized lesions on the limbs or trunk without distant metastases.
4. Experience primary tumor or local recurrence after surgery (disease-free survival more than 2 months after surgery)
5. Aged from 18 to 70, with ECOG performance status 0-1, or aged from 70 to 75, with ECOG performance status 0. Has life expectancy more than 2 years
6. Demonstrate adequate organ function (bone marrow, liver, and kidney function) (Leukocytes ≥ 3 × 10^9 /L, Neutrophils ≥ 1.5 × 10^9 /L, Hemoglobin ≥ 90 g/L, Platelet count ≥ 100 × 10^9 /L, Total bilirubin ≤1.5 × institutional upper limit of normal (ULN), Aspartate transaminase ≤2.5 × ULN, Alanine transaminase ≤2.5 × ULN, Serum creatinine ≤1.5 × ULN or creatinine clearance ≥60 mL/min.)
7. Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

1. The presences of regional or distant metastases detected by imaging evaluation
2. Patients with the following histological types: osteosarcoma, chordoma, classical chondrosarcoma, Kaposi's sarcoma, malignant mesothelioma, radiation-induced sarcomas.
3. Known history of another primary malignant tumor within the past three years or at the same time (excluding localized basal cell carcinoma, cutaneous squamous cell carcinoma, ductal carcinoma in situ, lobular carcinoma in situ, adenocarcinoma in situ of cervix, or other previous malignant tumor with a disease-free survival of more than five years)
4. Known history of other chemotherapy within 4 weeks before enrolment, previous anti-PD1 treatment, previous radiotherapy in the radiation field, or has other contraindications to radiotherapy or surgery.
5. Uncontrolled hyperglycaemia or Coagulation disorder
6. Active infection requiring systemic anti-infective therapy
7. Previous major surgery within 2 weeks before enrolment (excluding minor operation such as diagnostic biopsy or peripherally inserted central catheter implantation)
8. Known history of immunodeficiency diseases or active autoimmune disease requiring systemic treatment
9. Female patients pregnant or breastfeeding, Male patients expecting to have babies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2024-08-24 (Estimated); Study Completion 2029-08-24 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | The objective response rate (ORR) will be evaluated before surgery, which will be scheduled 5-12 weeks after the last fraction of radiotherapy.
  The percentage of patients with objective response. Objective response is defined as complete response (CR) or partial response (PR) per response evaluation criteria (RECIST v1.1) before surgery.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) and Near pCR Rate | The pathologic complete response (pCR) rate will be evaluated from surgical samples, immediately after surgery.
  The proportion of subjects whose pathological response rate of tumor tissue in postoperative specimens is ≥90% after preoperative treatment.
Non-Perfused Volume (NPV) | The non-perfused volume (NPV) will be measured in four weeks before preoperative treatment and before surgery, which will be scheduled 5-12 weeks after the last fraction of radiotherapy.
  The changes in tumour volume that are not enhanced in imaging images with contrast agent before and after treatment.
Acute Adverse Events | through study completion, an average of 6 months.
  The toxic reactions are evaluated and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Edition 5 (NCI-CTCAE V. 5).
Wound Complications | Up to 120 days from the surgery.
  Postoperative incision healing, with reference to the Canadian study for grading of wound complications.
Local Control Rate | Up to 5 years
  The proportion of subjects who recurred within the radiotherapy exposure field from initiation of treatment to the imaging assessment of all evaluable subjects.
Progression-Free Survival (PFS) | Up to 5 years
  The time from initiation of treatment to PD or death from any cause.
Overall Survival (OS) | Up to 5 years
  The time from initiation of treatment to death from any cause.
Quality of Life (QoL) according to the Musculoskeletal Tumor Society (MSTS) | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Musculoskeletal Tumor Society (MSTS) is a measure of physical function across 7 items, including pain, range of motion, strength, joint stability, joint deformity, emotional acceptance, and overall function. Each item is scored from 0(worst) to 5(best) with a maximum possible score of 35, which is converted to a scale from 0 to 100 points.
Quality of Life (QoL) according to the Toronto Extremity Salvage Score (TESS) | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Toronto Extremity Salvage Score (TESS) is a self-administered questionnaire evaluating possible limitations in physical activity. A total of 30 questions are included in the TESS, and the degree of disability is rated from 0 (complete disability) to 5 (no functional impairment) in each item.
Quality of Life (QoL) according to the Short Form (SF)-36 questionnaires | Quality of Life (QoL) will be evaluated at least five times: before treatment, at 3, 6, 12 and 24 months respectively after surgery.
  The Short Form (SF)-36 questionnaires is a 36-item health survey status which is composed of the following eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each of these domains can be rated from 0 (worst) to 100 (best). The final SF-36 score is converted to a 0-100 points range scale.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, M.D, PH.D, Principal Investigator — Fudan University; Wangjun Yan, M.D, PH.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China